CLINICAL TRIAL: NCT04276077
Title: Effects of Different Electrical Muscle Stimulation on Muscle Stiffness and Functional Capacity in Post-menopausal Women
Brief Title: Electrical Muscle Stimulation on Muscle Stiffness and Functional Capacity in Post-menopausal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, César Calvo Lobo, Principal Investigator, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMS_US
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Electric Stimulation Therapy; Frailty; Women
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-frequency electrical muscle stimulation (Experimental)
  Interventions: Other: High-frequency electrical muscle stimulation training
- Low-frequency electrical muscle stimulation (Experimental)
  Interventions: Other: Low-frequency electrical muscle stimulation training
- Control (No Intervention)

INTERVENTIONS:
Other: High-frequency electrical muscle stimulation training — High-frequency electrical muscle stimulation training with 50 Hertz during 8 weeks
  Arms: High-frequency electrical muscle stimulation
Other: Low-frequency electrical muscle stimulation training — Low-frequency electrical muscle stimulation training with 10 Hertz during 8 weeks
  Arms: Low-frequency electrical muscle stimulation

SUMMARY:
The aim of this study will be to determine the effects of different electrical muscle stimulation protocols on muscle stiffness and functional capacity in post-menopausal women. A randomized controlled clinical trial will be carried out. A total sample of 27 post-menopausal women will be recruited and divided into 3 groups which received high-frequency electrical muscle stimulation during 8 weeks, low-frequency electrical muscle stimulation during 8 weeks or no-intervention (control group). Outcome measurements will be stiffness assessed by sonoelastography and functional capacity assessed by the 30 seconds Chair-Stand Test before and after 8 weeks interventions.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women

Exclusion Criteria:

* Arrhythmias
* Diabetes
* Smokers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Stiffness | Change from Baseline stiffness at 8 weeks
  Quadriceps stiffness will be measured in Pascals by sonoelastography

SECONDARY OUTCOMES:
Functional capacity | Change from Baseline functional capacity at 8 weeks
  Functional capacity will be measured in repetitions by the 30 seconds Chair Stand Test

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Francisco de Vitoria, Pozuelo de Alarcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided